CLINICAL TRIAL: NCT05941481
Title: Neoadjuvant Chemo-hypofractionated Radiotherapy Plus PD-1 Antibody (Tislelizumab) in Locally Advanced Resectable Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Neoadjuvant Chemo-hypoRT Plus PD-1 Antibody (Tislelizumab) in Resectable LA-G/GEJ
Acronym: RARE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Cheng Chen, M.D, Jiangsu Cancer Institute & Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: jsCANCER
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Gastric or Gastroesophageal Junction Adenocarcinoma
Keywords: gastric or gastroesophageal junction adenocarcinoma; neoadjuvant chemo-hypofractionated radiotherapy; PD-1 Antibody
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- neoadjuvant chemo-hypofractionated radiotherapy plus PD-1 antibody (Experimental): 1. Immunotherapy combined with chemotherapy (2 cycles): Intravenous tislelizumab (200mg, d1, q21d) in combination with XELOX regimen (capecitabine 1000 mg/m2 bid*14d + oxaliplatin 130mg/m2, d1, q21d);
  2. Concurrent radiotherapy: Within one week after the first initiation of chemo-immunotherapy, concurrent hypofractionated radiotherapy will be started: intensity modulated radiotherapy was given for tumors, total dose:30Gy/12f, 2.5Gy/f.
  3. D2 resection will be received three to five weeks after the completion of neoadjuvant therapy.
  Interventions: Combination Product: neoadjuvant chemo-hypofractionated radiotherapy plus PD-1 antibody (Tislelizumab)

INTERVENTIONS:
Combination Product: neoadjuvant chemo-hypofractionated radiotherapy plus PD-1 antibody (Tislelizumab) — 1. Immunotherapy combined with chemotherapy (2 cycles): Intravenous tislelizumab (200mg, d1, q21d) in combination with XELOX regimen (capecitabine 1000 mg/m2 bid*14d + oxaliplatin 130mg/m2, d1, q21d);
  2. Concurrent radiotherapy: Within one week after the first initiation of chemo-immunotherapy, concurrent hypofractionated radiotherapy will be started: intensity modulated radiotherapy was given for tumors, total dose:30Gy/12f, 2.5Gy/f.

SUMMARY:
Gastric cancer is the third leading cause of death due to cancer worldwide. Although the consensus on the surgical treatment has resulted in the improvement of curative effect during the past decades, controversies remained for the perioperative therapy of gastric cancer, especially in the selection of the optimal neoadjuvant regimens. Immunotherapy with anti-programmed cell death-1 (PD-1) antibody has demonstrated moderate efficacy in selected patients with advanced gastric adenocarcinoma. Hypofractionated radiotherapy (HypoRT) may act synergistically with immunotherapy to enhance antitumor responses. This phase II trial study want to exploit the efficacy and safety to give PD-1 antibody (Tislelizumab) with combination chemotherapy and HypoRT before surgery in treating adult patients with gastric or gastroesophageal junction adenocarcinoma.

DETAILED DESCRIPTION:
1. This clinical trial will be conducted under Simon's optimal two-stage design. The first stage needs 9 participants, if ≥1 participants acquire remission, then the study will move on to the second stage and enroll the rest 10 participants. Taking into account a drop-out rate of about 5%, we planned to enroll 21 patients.
2. Target population: patients with resectable locally advanced resectable gastric or gastroesophageal junction adenocarcinoma (cT1-2N+M0/T3-T4aNanyM0).
3. Trial design: This is a monocenter, single arm, phase II study to evaluate the efficacy and safety of neoadjuvant chemo-hypofractionated radiotherapy plus PD-1 antibody (Tislelizumab) in patients with locally advanced gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma involving the gastroesophageal junction or gastric cardia.
2. Having an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 within 7 days before enrollment.
3. Being histologically diagnosed with adenocarcinoma.
4. Having tumor lesions at stomach or gastroesophageal junction (Siewert type II or III);
5. Clinically diagnosed stage T1-2N+M0/T3-T4aNanyM0 according to ultrasound endoscopy or enhanced CT/MRI scan.
6. At least one evaluable lesion in abdominal CT/MRI according to RESIST 1.1 is required.
7. Surgical consultation at enrolling site to confirm that patient will be able to undergo curative resection after completion of neoadjuvant therapy =< 56 days prior to registration.
8. Physical condition and adequate organ function to ensure the success of abdominal surgery.
9. Adequate hematological function: Neutrophil count ≥ 1.5 × 109/L, Platelets ≥ 100 × 109/L and Hemoglobin ≥90g/L.
10. Adequate liver function: Total bilirubin ≤ 1.5 × upper limit of normal (ULN); AST (SGOT) and ALT (SGPT) < 2.5 × ULN in the absence of liver metastases, or < 5 × ULN in case of liver metastases. ALP ≤ 2.5 × upper limit of normal (ULN); ALB ≥30g/L.
11. Adequate renal function: Serum creatinine ≤ 1.5 x ULN, and creatinine clearance ≥ 60 ml/min.
12. Adequate coagulation function: INR/PT≤ 1.5 x ULN, aPTT≤ 1.5 x ULN.
13. No serious concomitant disease that will threaten the survival of patients to less than 5 years.
14. Male or female. Age ≥ 18 years and ≤80 years.
15. Written (signed) informed consent.
16. Good compliance with the study procedures, including lab and auxiliary examination and treatment.
17. Female patients should not be pregnant or breast feeding.
18. Female patients of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication.

Exclusion Criteria:

1. Patients with distant metastasis or unresectable primary lesion.
2. Received prior treatment or receiving current treatment for this malignancy.
3. Patients who have digestive tract bleeding in 2 weeks before recruitment or with high risk of bleeding.
4. Perforation / fistula of GI tract in 6 months before recruitment.
5. Patients with upper GI tract obstruction or functional abnormality or malabsorption syndrome, which can affect absorption of apecitabine.
6. Patients with active autoimmune disease or history of refractory autoimmune disease.
7. Patients with active malignant tumor in recent 2 years, except the tumor studied in this research or cured locally tumor like resected basal cell or squamous cell skin cancer, superficial bladder cancer, cervical or breast carcinoma in situ.
8. Uncontrollable pleural effusion, pericardial effusion, or ascites in 2 weeks before recruitment.
9. Pulmonary disease history: interstitial pulmonary disease, non-infective pneumonitis, pulmonary fibrosis, acute pulmonary disease.
10. Uncontrollable systemic diseases, including diabetes, hypertension, etc.
11. Severe chronic or active infections in need of systemic antibacterial, antifungal, or antiviral treatment, including TB or HIV, etc.
12. Patients with untreated chronic hepatitis B or HBV DNA over 500 IU/ml or positive HCV RNA.
13. Patients with any cardiovascular risk factors below:

    1. cardiac chest pain occurring in 28 days before recruitment, defined as moderate pain that limits daily activity.
    2. pulmonary embolism with symptoms occurring in 28 days before recruitment.
    3. acute myocardial infarction occurring in 6 months before recruitment.
    4. any history of heart failure reaching grade 3/4 of NYHA in 6 months before recruitment.
    5. ventricular arrhythmias of Grade 2 or grater in 6 months before recruitment, or accompanied by supraventricular tachyarrhythmias requiring medical treatment.
    6. cerebrovascular accident within 6 months before recruitment.
14. Moderate or severe renal injury [creatinine clearance rate≤50 ml/min (according to Cockroft & Gault equation)], or Scr>ULN.
15. Dipyrimidine dehydrogenase (DPD) deficiency.
16. Allergic to any drug in this study.
17. History of allogeneic stem cell transplantation or organ transplantation.
18. Use of steroids (dosage>10mg/d prednisone) or other systemic immune suppressive therapy in 14 days before recruitment, except patients treated with regimens below: a. steroids for hormone replacement (dosage>10mg/d prednisone); b. steroids for local application with little systemic absorption; c. short -term (≤ 7 days) steroids for preventing allergy or vomiting.
19. Vaccinated with live vaccine in 4 weeks before recruitment.
20. Receiving immune (interleukin, interferon, thymin) treatment or treatment of other trials in 28 days before recruitment.
21. Receiving palliative radiation in 14 days before recruitment.
22. History of anti PD-1, PD-L1, PD-L2 or any other specific T cell co-stimulation or checkpoint pathway targeted treatment.
23. Patients who lose ≥20% of body weight within 2 months before enrollment.
24. For patients with uncontrolled epilepsy, CNS diseases or history of mental disorder, researchers should evaluate whether their diseases will impede their signing of informed consent or compliance of treatment.
25. Existing of potential situation which will impede drug administration or affect toxicity analysis or alcohol/ drug abuse.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-06-10 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
pathological complete remission (pCR) rate | From date of treatment allocation and during treatment period up to 1 year
  Pathologic complete response was defined as pT0N0M0

SECONDARY OUTCOMES:
Radiographic response | From date of treatment allocation and during treatment period up to 3 months
  To assess radiographic response to neoadjuvant tislelizumab with concurrent chemoradiotherapy using RECIST 1.1.
The R0 resection rate | Up to 3 years
  Complete Resection With no Tumor Within 1 mm of the Resection Margins (R0) Rate
Safety of neoadjuvant chemo-hypofractionated radiotherapy plus PD-1 antibody (Tislelizumab) Safety of neoadjuvant therapy | 1 month after the last date of treatment
  Adverse events (AE) of neoadjuvant therapy will be graded and documented according to NCI-CTCAE v5.0 from the beginning of treatment to 1 month after the last date of treatment.
Postoperative complications | AEs of surgery refer to complications which happen during or in 30 days after operation.
  Using the Clavien-Dindo classification
Time to Relapse (TTR) | Time from the date of study registration to the date of 1st documented relapse/recurrence among patients who achieve R- resection, assessed up to 3 years
  The median TTR and confidence interval will be estimated using the method of Kaplan-Meier
Progression-free Survival (PFS) | Time from the date of study registration to the date of death due to all causes, recurrences if R0 resections are achieved, progression disease before undergoing surgery, or R1/R2 resection at surgery, whichever comes first, assessed up to 3 years
  The distribution of PFS will be estimated using the method of Kaplan-Meier.
Overall Survival (OS) | Time from the date of study registration to the date of death due to all causes, assessed up to 3 years
  The distribution of OS will be estimated using the method of Kaplan-Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Chen, doctor, Principal Investigator — Jiangsu Cancer Institute & Hospital
Locations (1):
- Jiangsu Cancer Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No